CLINICAL TRIAL: NCT00399880
Title: Improving Medication Adherence Through Graphically Enhanced Interventions in Acute Coronary Syndromes
Acronym: IMAGE-ACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Society of Health-System Pharmacists Research and Education Foundation (Other)
Responsible Party: Principal Investigator, Sunil Kripalani, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00000116; K23HL077597 (NIH)
Record Dates: First submitted 2006-11-13; First posted 2006-11-15 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-07

CONDITIONS: Acute Coronary Syndrome (ACS)
Keywords: Clinical Trial; Behavioral/Social; Cardiovascular Disease; Risk Factors/Analysis
MeSH Terms: conditions — Acute Coronary Syndrome; Behavior; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health literacy intervention (Experimental): Illustrated medication schedules, pill boxes, pharmacist counseling
  Interventions: Behavioral: Health literacy intervention
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Health literacy intervention — Illustrated medication schedules, pill boxes, pharmacist counseling
  Arms: Health literacy intervention

SUMMARY:
Coronary heart disease (CHD) is the leading cause of death in the United States. Most people who die from CHD die of a heart attack. Acute coronary syndrome (ACS) is a term that includes mild heart attacks, as well as other episodes of chest pain that may serve as a warning sign for an upcoming heart attack.

There are many medicines that can help prevent and treat ACS. However, at least 25% of patients don't take their medications as prescribed. When patients don't take their medications, we say they are noncompliant or nonadherent with the treatment.

The period following hospital discharge is a vulnerable time for many patients. Patients are often confused about what to do when they return home from the hospital. Many patients don't take their medications correctly, or they don't take them at all. Patients with poor literacy skills have more trouble than others, because it is harder for them to follow written instructions. Overall, about half of the adults in the U.S. have poor literacy skills. It is important to develop ways to help these adults manage their health better.

The purposes of this research project are 1) to learn more about the relationship between low literacy and medication adherence after hospital discharge, and 2) to test a strategy designed to help patients take their medicines more regularly. We will recruit consenting patients hospitalized with ACS. We will measure their literacy skills, ask questions about how they take their medicines, and measure other related factors like social support and self-efficacy. Patients will then be assigned to 1 of 2 groups. One group will receive only usual care at hospital discharge, which usually includes the nurse and physician briefly reviewing the medication prescriptions. The other group will receive an illustrated daily medication schedule and special, tailored counseling from a pharmacist at their time of discharge. About 1 week after patients leave the hospital we will contact them by phone to ask them questions about how they have been taking their medicines. We will get data from patients records for 6 months to see if the intervention had an impact on their medication compliance, blood pressure, cholesterol, and diabetes measurements.

If this study is successful, this simple strategy could be implemented by hospitals to improve medication compliance after discharge. This study will also provide more information about how patients' literacy skills affect their medication compliance.

ELIGIBILITY:
Inclusion Criteria:

- Present with acute chest pain or angina equivalent, lasting ≥ 10 minutes of suspected ischemic origin, within the previous 24 hours of presentation to the hospital.

PLUS

* Patient must have documented objective evidence of myocardial ischemia based on a or b:

  1. EKG changes in ≥ 2 contiguous leads shown by:

     * Transient (< 30 min) ST-segment elevation of ≥ 1.0mm

     OR

     * Transient or persistent ST-segment depression of ≥ 0.5mm (flat or downsloping at the J-point and at 80ms after the J-point)

     OR

     * Persistent T-wave inversion of ≥ 2.0mm
  2. Abnormal elevation of cardiac enzymes

     * Elevation of creating kinase (CK) and creatine kinase-myocardial band (CK-MB)

     OR

     * Elevation of troponin

     Exclusion Criteria:
* Previously enrolled in the study
* Police custody
* Corrected visual acuity worse than 20/60
* Lack of cooperation
* Severe hearing impairment
* Too ill to participate
* Unintelligible speech
* Age younger than 18 years
* Native language other than English
* Psychotic illness
* Caregiver administers all medications
* Delirium/severe dementia
* Does not fill prescriptions at Grady
* No regular telephone/address
* Not taking chronic medications prior to admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Kripalani, MD, MSc, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Usual care arm
Period: Overall Study
Arm/Group | Health Literacy Intervention | Usual Care
Started | 65 | 65
Completed | 65 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Literacy Intervention | Usual Care | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (9.2) | 52.2 (10.7) | 52.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 56
  Male | 38 | 36 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 62 | 63 | 125
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Income [Count of Participants; unit: Participants]
  <$10,000 | 40 | 44 | 84
  $10,000-$20,000 | 18 | 12 | 30
  >$20,000 | 5 | 5 | 10
  Missing | 2 | 4 | 6
Employment status [Count of Participants; unit: Participants]
  Unemployed | 31 | 20 | 51
  Full-time | 5 | 4 | 9
  Part-time | 3 | 4 | 7
  Other (disabled, retired) | 24 | 36 | 60
  Missing | 2 | 1 | 3
Education [Mean (Standard Deviation); unit: years] | 11.6 (3.0) | 11.5 (2.9) | 11.6 (2.9)
Rapid Estimate of Adult Literacy in Medicine (REALM) [Mean (Standard Deviation); unit: units on a scale] — Validated measure of health literacy involving participants' ability to read medical terms from a list. Possible range of scores 0-66, with higher values indicating better literacy.
  units on a scale | 41.1 (21.7) | 39.1 (22.7) | 40.1 (22.1)
Smoking status [Count of Participants; unit: Participants]
  Never | 18 | 29 | 47
  Former | 14 | 5 | 19
  Current | 33 | 28 | 61
  Missing | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Refills and Medications Scale (ARMS)
Description: Validated self-report measure of medication adherence. Possible range 12-48, with lower values indicating better adherence.
Time Frame: Approximately 2 weeks after hospital discharge
Population: Participants who were able to be contacted and provided outcome data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health Literacy Intervention | Usual Care
Number analyzed (Participants) | 38 | 38
units on a scale | 12.03 (2.59) | 12.18 (3.81)

2. Secondary Outcome: Self-Efficacy for Appropriate Medication Use Scale (SEAMS)
Description: Validated measure of confidence in taking medications correctly. Possible range 13-39, with higher values indicating greater confidence.
Time Frame: Approximately 2 weeks after hospital discharge
Population: Participants who were able to be contacted and provided outcome data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Health Literacy Intervention | Usual Care
Number analyzed (Participants) | 39 | 42
units on a scale | 32.8 (4.8) | 31.5 (6.7)

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- Usual Care: Usual care (Standard)
Arm/Group | Health Literacy Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 0/65 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No